CLINICAL TRIAL: NCT04223973
Title: Demonstration Study of the Interest of the MEDTRUM A7+ TouchCare Insulin Patch Pump Versus INSULET Omnipod® Patch Pump
Brief Title: MEDTRUM A7+ TouchCare Insulin Patch Pump (MedInPS)
Acronym: MedInPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtrum France (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-A02566-51
Record Dates: First submitted 2019-12-11; First posted 2020-01-13 (Actual); Results first posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus
Keywords: diabetes management; Insulin Pump
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (RCT), open-label with two arms, multicentric national, prospective, non-inferiority methodology versus reimbursed comparator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Group (Experimental): Using the Medtrum Pump A7+ during 3 months
  Interventions: Device: Medtrum A7+ insulin Pump; Biological: Lab A1C
- Control Group (Active Comparator): using the usual Insulet Patch pump
  Interventions: Biological: Lab A1C

INTERVENTIONS:
Device: Medtrum A7+ insulin Pump — Use of the Medtrum pump during 3 months in combination with a CGM (Continuous Glucose Measurement)
  Arms: Active Group
Biological: Lab A1C — Measure of Lab A1C at baseline and end of study

SUMMARY:
Demonstration study of the interest of the MEDTRUM A7+ TouchCare insulin patch pump versus INSULET Omnipod® patch pump

DETAILED DESCRIPTION:
Compare the daily use of two single usage patch pumps and demonstrate the interest of use of the A7+TouchCare® (Medtrum) patch pump for type 1 & 2 diabetes management.

Main objective is an estimation of Patients A1C (Glycated Haemoglobin) based on the average blood glucose (obtained from a Flash glucose monitoring) and to compare it in both groups.

Secondary objectives:

* comparison of mean A1C (laboratory values) between the two groups at Baseline and study end. Comparison to be established in a non-inferiority
* Observe Skin & overall Tolerance, Technical incidents with the device (failure, disconnection, catheter obstruction…)
* Collection of Glucose metrics (minimum, maximum, average/median, standard deviation, out of range value, percentage of time in range, glucose variability)

ELIGIBILITY:
Inclusion Criteria:

* Patient with type 1 or 2 diabetes, 18 years of age and over
* Patients already equipped with Omnipod® ® (INSULET) insulin patch pump and Abbott FreeStyleLibre sensor®.
* A1C ranking from : >= 6,5% to <= 9.5%
* Any type of rapid insulin except FIASP (which can be substituted if necessary) with 60 IU max per day (unauthorized use of insulin supplements by pen injector)
* Patient able to receive and understand study information, give written informed consent, and easily participate to the trial
* Patient affiliated to the French social security system

Exclusion Criteria:

* - Patient already participating in another study
* Patient under the protection of justice or under guardianship or curatorship
* Type 2 diabetic patient requiring a daily insulin dose > 60 IU
* Patients not suitable for suing insulin pump such as: severe psychiatric disorders, rapidly progressing ischemic or proliferative retinopathy before laser treatment, and exposure to high magnetic ﬁelds
* Patients allergic to nickel and adhesive
* Pregnant women, breastfeeding women
* Or any other criteria as appreciated by the study investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Freddy PENFORNIS, Principal Investigator — Centre Hospitalier Francilien, Corbeil
Locations (1):
- Centre hospitalier Sud Francilien, Corbeil-Essonnes, Essones, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amadou C, Melki V, Allain J, Clavel S, Gouet D, Chaillous L, Catargi B, Schaeplynck-Belicard P, Petit C, Thivolet C, Penfornis A. Performance and patients' satisfaction with the A7+TouchCare insulin patch pump system: A randomized controlled non-inferiority study. PLoS One. 2023 Aug 24;18(8):e0289684. doi: 10.1371/journal.pone.0289684. eCollection 2023. PMID 37616289

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of recruitment: January 2020 to February 2021 > total duration 13 months 8 investigational centres mainly hospitals (General and University Hospitals)
Pre-assignment Details: Due to Covid 19 pandemia some clinical sites Research Department decided to stop recruitment or put interventional arm of the protocol of test on hold. As consequence of this, some participants where withdrawn. Mainly in Active group as in the control group patients were using their usual devices and treatment and they resumes follow up visits as usual.
Groups:
- Medtrum A7+ Insulin Pump: Using the Medtrum Pump A7+ during 3 months
  Medtrum A7+ insulin Pump: Use of the Medtrum pump during 3 months in combination with a CGM
  Lab A1C: Measure of Lab A1C at baseline and end of study
- Insulet Patch Pump: Patients using their usual device: Insulet Patch pump
  Lab A1C: Measure of Lab A1C at baseline and end of study Use of their usual pomp and usual CGM during 3 months
Period: Overall Study
Arm/Group | Medtrum A7+ Insulin Pump | Insulet Patch Pump
Started | 48 | 45
Completed | 35 | 43
Not Completed | 13 | 2
Not completed — Patients 'withdrawal due to Covid 19 impact on study recruitment/follow-up on site | 5 | 0
Not completed — Adverse Event | 4 | 0
Not completed — patients reported product dysfunctions and decided to stop the study | 3 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Per protocol population (78 participants)
Groups:
- Medtrum A7+ Insulin Pump: Patients use the Medtrum A7+ insulin Pump during 3 months in combination with a Continuous Glucose Monitoring (CGM)
- Insulet Patch Pump: Patients carry on using their usual Insulet Patch pump in combination with a CGM
- Total: Total of all reporting groups
Arm/Group | Medtrum A7+ Insulin Pump | Insulet Patch Pump | Total
Number analyzed (Participants) | 48 | 45 | 93
Age, Customized [Mean (Standard Deviation); unit: years] — Measures at baseline were collected in a Case report form and check with Patient medical record
  years
    Population age | 49.4 (11.7) | 50.3 (13.6) | 49.8 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 29 | 53
  Male | 24 | 16 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI (kg/m²) [Mean (Standard Deviation); unit: kg/m^2] | 26.5 (4.1) | 25.4 (4.3) | 26.0 (4.2)
Diabetes type [Count of Participants; unit: Participants]
  Type 1 diabetics | 41 | 43 | 84
  Type 2 diabetics | 7 | 2 | 9
Time since diabetes diagnosis [Mean (Standard Deviation); unit: years] | 22.7 (11.1) | 22.2 (11.5) | 22.5 (11.3)
Time since initiation of insulin pump treatment [Mean (Standard Deviation); unit: years] | 5.4 (4.3) | 7.1 (6.7) | 6.2 (5.7)
A1C measured at lab Vs sensor estimation [Mean (Standard Deviation); unit: percentage of hemoglobin A1C]
  Laboratory A1C | 7.8 (0.7) | 7.8 (0.8) | 7.8 (0.7)
  Sensor estimated A1C | 7.5 (0.9) | 7.4 (0.8) | 7.4 (0.9)
Insulin /day [Mean (Standard Deviation); unit: IU/day]
  Daily basal dose | 18.7 (10.0) | 16.1 (5.9) | 17.5 (8.4)
  Daily Bolus Dose | 18.7 (10.9) | 21.5 (9) | 20 (10.1)

OUTCOME MEASURES:

1. Primary Outcome: Estimation of A1C (%) Based on Average Blood Glucose Measured by Continuous Glucose Sensor on the Last 10 Weeks
Description: A1C will be estimated by a Continuous Glucose Measurement (FreeStyle Libre®) for all patients, at baseline and end of the study (12 weeks). The main objective is to demonstrate Non-inferiority efficacy (PP then ITT) of Medtrum A7+ insulin patch pump vs Insulet Omnipod® insulin patch pump (2 randomized groups). For the primary outcome, A1C will be estimated and appear in percentage based on assessment done by a Continuous Glucose Monitoring system.
  The A1C obtained in real life for the group using the comparator pump (Omnipod®) is estimated at 7.8%. Assuming that blood glucose level will be the same with Medtrum pump and based on a defined non-inferiority margin ∆ = + 0.4 (following FDA Guidance for Industry Diabetes Mellitus: Developing Drugs and Therapeutic Biologics for Treatment and Prevention).
Time Frame: Month 3
Population: population analysed is population per protocol: population wearing the sensor and using the pump at least 90% of time over the last 10 weeks of protocol (out of 12 weeks total study duration)
Measure: Least Squares Mean (Standard Deviation); unit: estimated percentage of hemoglobin A1C
Groups:
- Medtrum A7+ Insulin Pump: Patients Using the Medtrum A7+ insulin Pump during 3 months in combination with a CGM
  Lab A1C: Measure of Lab A1C at baseline and end of study
- Insulet Patch Pump: Patients using their usual Insulet Patch pump in combination with a CGM
  Lab A1C: Measure of Lab A1C at baseline and end of study
Arm/Group | Medtrum A7+ Insulin Pump | Insulet Patch Pump
Number analyzed (Participants) | 35 | 43
estimated percentage of hemoglobin A1C | 7.345 (0.094) | 7.347 (0.085)

2. Secondary Outcome: Report Patients' Laboratory Hemoglobin A1C Difference Between Baseline and 3 Months
Description: A1C is expressed in percentage based on Laboratory measurement. A1C is obtained & measured from a blood sample.
Time Frame: Month 3
Population: population per protocol as population wearing their sensor 90% of time and wearing their pump 90% of time over the last 10 weeks of the test duration
Measure: Mean (Standard Deviation); unit: percentage of laboratory hemoglobin A1C
Groups:
- Medtrum A7+ Insulin Pump: Patient using the Medtrum A7+ insulin Pump during 3 months in combination with a CGM
- Insulet Patch Pump: Patients using their usual Insulet Patch pump in combination with their usual CGM
Arm/Group | Medtrum A7+ Insulin Pump | Insulet Patch Pump
Number analyzed (Participants) | 35 | 43
percentage of laboratory hemoglobin A1C | -0.057 (0.475) | 0.007 (0.496)

3. Secondary Outcome: Compare The Time Spent in Range
Description: Glycemic Time In Range is the Time spent in the target. It is expressed in % of time.
  Time in Range is automatically calculated from the Sensor data wear.
Time Frame: Month 3
Population: Modified Intent-To-Treat population (ITTm) as population with FSL (FreeStyle Libre) available data at 3 months
Measure: Mean (Standard Deviation); unit: percentage of time spent in the target
Groups:
- Medtrum A7+ Insulin Pump: Patients using the Medtrum A7+ insulin Pump during 3 months in combination with a CGM
- Insulet Patch Pump: Patients using their usual insulin pump in combination with a CGM during 3 months
Arm/Group | Medtrum A7+ Insulin Pump | Insulet Patch Pump
Number analyzed (Participants) | 36 | 43
percentage of time spent in the target | 56.5 (12.3) | 58.4 (13.1)

4. Secondary Outcome: Compare Patients Pump Satisfaction
Description: Question: Overall, how satisfied were you with the pump? Satisfaction to be measured by a Patient Self- questionnaire through a Likert scale ranking from 1 (the less) to 5 (the most).
Time Frame: Month 3
Population: population ITTm as population with available questionnaire data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medtrum A7+ Insulin Pump | Insulet Patch Pump
Number analyzed (Participants) | 36 | 43
units on a scale | 3.5 (1.2) | 4.1 (0.7)

5. Secondary Outcome: Compare Patients PDM Satisfaction
Description: Question: How to qualify the discretion of use of the PDM (Personal Diabetes Manager) of the pump? the satisfaction scale went from 1 (very unsatisfied) to 5 (very satisfied)
Time Frame: Month 3
Population: population ITTm as population with available questionnaire data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Medtrum A7+ Insulin Pump | Insulet Patch Pump
Number analyzed (Participants) | 36 | 43
units on a scale | 4.4 (0.8) | 3.8 (1.0)

6. Secondary Outcome: Number of Participants With at Least One Pump Occlusion
Description: occlusion reported by patient
Time Frame: Month 3
Population: population ITTm as population with available questionnaire data
Measure: Count of Participants; unit: Participants
Arm/Group | Medtrum A7+ Insulin Pump | Insulet Patch Pump
Number analyzed (Participants) | 36 | 43
Participants | 24 | 12

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Medtrum A7+ Insulin Pump | Insulet Patch Pump
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/45
Serious Adverse Events (participants affected / at risk) | 1/48 | 0/45
Other Adverse Events (participants affected / at risk) | 7/48 | 2/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medtrum A7+ Insulin Pump (N=48) | Insulet Patch Pump (N=45)
Ketonemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medtrum A7+ Insulin Pump (N=48) | Insulet Patch Pump (N=45)
Bleeding at the injection site (General disorders) | 4 (4) | 2 (2)
Pain at the injection site (General disorders) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
15 patients were excluded from the PP Population due to protocol deviations (mainly premature discontinuation due to COVID 19 context), which occurred more frequently in the Touchcare group (13 patients vs 2 patients in the Omnipod group).

Some differences in favour of the Omnipod pump may be explained since patients in this group used the Omnipod pump (and already satisfied with it) since several months or years, compared to only 1 to 3 months of use with the unknown Touchcare pump.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/73/NCT04223973/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/73/NCT04223973/SAP_001.pdf